CLINICAL TRIAL: NCT01780402
Title: Comparison of Hand Feeding Techniques for Persons With Dementia Living in the Nursing Home
Brief Title: Comparison of Hand Feeding Techniques for Persons With Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: The John A. Hartford Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Supportive Care
Other Study IDs: Pro00035130
Record Dates: First submitted 2013-01-29; First posted 2013-01-31 (Estimated); Last update posted 2016-10-06 (Estimated); Status verified 2016-10

CONDITIONS: Dementia
Keywords: feeding difficulty; eating difficulty; dementia; nursing home; careful hand feeding
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Hand feeding intervention delivery (Experimental): Trained Research Feeding Assistants (TRFA), blind to the study outcomes, will assist enrolled PWDs with all three meals for two days using a pre-specified hand feeding technique. Videotaping will occur for two enrolled PWD during the six day time frame to promote efficiency. Coding of the video will be done by a trained Data Technician after meals have been recorded to determine frequency of aversive feeding behaviors, calculate meal intake, and time spent assisting with the meal.
  Interventions: Behavioral: Hand feeding techniques

INTERVENTIONS:
Behavioral: Hand feeding techniques — Direct hand feeding technique: When the feeding assistant holds the object (e.g., fork, spoon, cup) intended to provide food or fluids to the PWD without any active involvement on the part of the PWD.
  Hand-over-hand feeding technique: Occurs when the PWD is holding the object (e.g., fork, spoon, cup) in an attempt to feed/ drink for themselves. If the PWD has trouble with this activity, the feeding assistant puts his or her hand over the hand of the PWD, in an effort to guide/ support/ assist the PWD with the activity.
  Hand-under-hand feeding technique: Occurs when the feeding assistant holds the object (e.g., fork, spoon, cup) and places the PWD hand over the top of their hand; therefore, the feeding assistants hand is under the hand of the PWD in a more supportive position.
  Other Names: Direct hand feeding, hand over hand feeding, and hand under hand feeding.

SUMMARY:
The purpose of this study is to test three hand feeding techniques that can be used to provide feeding assistance to persons with dementia - direct hand feeding, hand-over-hand feeding, and hand-under-hand feeding.

DETAILED DESCRIPTION:
Proposed Aim 1: To collect pilot data related to using three hand feeding techniques for feeding persons with dementia (PWD) in the nursing home (NH) setting: (1) direct hand feeding; (2) hand-over-hand feeding; and, (3) hand-under-hand feeding. Primary outcomes are impact on frequency of aversive feeding behaviors, meal intake, and time spent assisting with feeding.

Proposed Aim 2: Evaluate implementation of the hand feeding intervention for larger randomized study of feeding techniques.

Aim 2a: Conduct a process evaluation for method of recruiting, screening, and obtaining informed consent of legally authorized representatives (LARs)/ assent of PWD.

Aim 2b: Establish fidelity to treatment for all three hand feeding interventions.

ELIGIBILITY:
Inclusion Criteria:

* Resident of nursing home 6 weeks prior to intervention delivery
* 60+ years old
* Have a legally authorized representative to provide informed consent
* medical diagnosis of dementia
* required extensive assistance to total dependence for feeding
* Brief Interview for Mental Status (BIMS) score of 0-12

Exclusion Criteria:

* Positive diagnosis of Human Immunodeficiency Virus (HIV), Parkinson's, and/or Traumatic Brain Injury
* Any swallowing disorder
* Presence of feeding tube that is sole source for meal delivery
* Significant auditory or visual impairment

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-03; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Change in frequency of aversive feeding behaviors | Day 6
  Changes in behaviors of person with dementia being assisted with 3 meals daily over 6 days
Changes in time spent providing feeding assistance | Day 6
  Changes in time spent providing feeding assistance to a person with dementia being assisted with 3 meals daily over 6 days
Changes in meal intake | Day 6
  Changes in meal intake for a person with dementia being assisted with 3 meals daily over 6 days

SECONDARY OUTCOMES:
Functional ability and feeding behaviors exhibited by person with dementia | Day 6
  Coding of video recorded meals from Outcomes 1-3
Characterize feeding assistant responses to functional ability and feeding behaviors | 6 days
  Coding of video recorded meals from Outcomes 1-3
Develop decision-making algorithm of adaptive approaches used by feeding assistant | 6 days
  Coding of video recorded meals from Outcomes 1-3

CONTACTS AND LOCATIONS:
Overall Officials: Melissa B Aselage, PhD,RN,FNP, Principal Investigator — Duke University School of Nursing; Ruth Anderson, PhD,RN,FAAN, Study Chair — Duke University School of Nursing; Elaine J Amella, PhD,RN,FAAN, Study Chair — Medical University of South Carolina
Locations (11):
- United States (11):
  - Rex Apex, Apex, North Carolina
  - Carolina Meadows, Chapel Hill, North Carolina
  - Carver Living Center, Durham, North Carolina
  - Croasdaile, Durham, North Carolina
  - Hillcrest, Durham, North Carolina
  - Pettigrew, Durham, North Carolina
  - Treyburn, Durham, North Carolina
  - Kindred Cypress Pointe, Wilmington, North Carolina
  - Wilmington Health & Rehabilitation Center, Wilmington, North Carolina
  - Liberty Commons Nursing Center, Wilmington, North Carolina
  - Davis Health Care Center, Wilmington, North Carolina

IPD SHARING:
Plan to Share IPD: Undecided